CLINICAL TRIAL: NCT02462590
Title: Probiotics to Prevent Severe Pneumonia and Endotracheal Colonization Trial (PROSPECT)
Brief Title: Probiotics to Prevent Severe Pneumonia and Endotracheal Colonization Trial
Acronym: PROSPECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27022015
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2019-01

CONDITIONS: Ventilator Associated Pneumonia; Infections; C-Difficile; Antibiotic-associated Diarrhea; Diarrhea
Keywords: Probiotics; Ventilator Associated Pneumonia; Infections; C-Difficile; Antibiotic-associated Diarrhea; Diarrhea
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus rhamnosus GG (Active Comparator): Patients allocated to the intervention group will receive 1x1010 colony forming units (CFU) of L. rhamnosus GG (Culturelle, Locin Industries Ltd) in 1 capsule suspended in tap water, administered through a nasogastric (or orogastric) or nasoduodenal (or oroduodenal) tube twice daily while patients are in the ICU. The first dose will be within 72 hours of intubation. Patients in the ICU who await discharge and can swallow pills will take the capsules orally.
  Interventions: Drug: L. rhamnosus GG - Probiotic
- Placebo (Placebo Comparator): Patients allocated to the placebo group will receive a capsule identical in appearance to the L. rhamnosus GG capsule, but containing microcrystalline cellulose. The placebo will also be suspended in tap water and similarly administered twice a day. When suspended in water, the placebo has identical appearance and consistency as the probiotic. The placebo will be prepared by the manufacturer of L. rhamnosus GG, Culturelle, and has been used successfully in a recent RCT in the ICU population [Morrow 2010]. This has also been used successfully in the PROSPECT Pilot Trial.
  Interventions: Drug: Placebo - Microcrystalline Cellulose

INTERVENTIONS:
Drug: L. rhamnosus GG - Probiotic — Twice daily, patients will receive either 1x1010 colony forming units (CFU) of L. rhamnosus GG (Culturelle, Locin Industries Ltd) in 1 capsule or an identical placebo capsule
  Other Names: Culturelle Probiotic
  Arms: Lactobacillus rhamnosus GG
Drug: Placebo - Microcrystalline Cellulose — Microcrystalline Cellulose
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Probiotics are commercially available live bacteria thought to have health benefits when ingested. A literature review of probiotic studies in the intensive care unit (ICU) found that in patients who receive probiotics, there is a 25% reduction in lung infection, known as ventilator-associated pneumonia (VAP). There is also an 18% reduction in the chance of developing any infection in the ICU. However, the studies reviewed were small and not well done. Therefore, whether probiotics are really helpful or not is unclear. Before a large carefully performed study is done to evaluate the effects of probiotics in critically ill patients, a pilot trial was needed. The Investigators completed a multicenter pilot RCT for which the primary outcomes relate to feasibility. Feasibility goals were met. 1) Recruitment for the Pilot was achieved in 1 year; 2) Adherence to the protocol was 96%; 3) There were no cases of contamination; 4) The VAP rate was 15%. This study is very important in the ongoing search for more effective strategies to prevent serious infection during critical illness. Probiotics may be an easy-to-use, readily available, inexpensive approach to help future critically ill patients around the world.

DETAILED DESCRIPTION:
Background:Probiotics are live microorganisms thought to have health benefits when ingested. Randomized controlled trials (RCTs) have documented favourable impact on a range of clinical problems, including prevention of upper respiratory tract infections, antibiotic-associated diarrhea, Clostridium difficile-associated diarrhea, and irritable bowel syndrome. Our recent meta-analysis of probiotic RCTs in the intensive care unit (ICU) also suggests 25% lower rates of ventilator-associated pneumonia (VAP) and 18% lower infection rates overall when administered to critically ill mechanically ventilated patients. However, these estimates arise from small, modest quality single-center RCTs yielding imprecise estimates of effect and uncertain generalizability, and require confirmation in a large methodologically rigourous RCT. Before launching a complex costly RCT testing whether probiotics confer benefit, harm, or have no impact on infectious and non-infectious outcomes, a pilot trial was needed. The investigators completed a multicenter pilot RCT for which the primary outcomes relate to feasibility: 1) recruitment success in 1 year; 2) >90% adherence to the probiotic protocol; 3) <5% contamination; 4) an estimated VAP rate. Patients have been randomized in 14 centers in Canada and the US, with an informed consent rate of 84%. Feasibility goals were met. 1) Recruitment for the Pilot was achieved in 1 year; 2) Adherence to the protocol was 96%; 3) There were no cases of contamination; 4) The VAP rate was 15%. This will be an internal Pilot which will be incorporated into the main trial.

Setting: 13 ICUs in Canada, 2 ICUs in United States

Methods: Patients age 18 years or older, admitted to the ICU, with an anticipated duration of ventilation of ≥72 hours are included. Patients are excluded if they have increased risk of iatrogenic probiotic infection or endovascular infection, primary diagnosis of severe acute pancreatitis, percutaneous gastric or jejunal feeding tubes already in situe, strict contraindication or inability to receive enteral medications, have hopeless prognosis, withholding or withdrawal of advanced life support is planned, or if previous enrolment in this or a related trial. Following informed consent, patients are randomized in variable unspecified block sizes in a fixed allocation ratio of 1:1, stratified by ICU and medical/surgical/trauma status. Twice daily, patients receive either 1x1010 colony forming units (CFU) of L. rhamnosus GG (Culturelle, Locin Industries Ltd) in 1 capsule or an identical placebo capsule. Both are suspended in water administered via nasogastric tube or by capsule. Research Nurses notify local Study Pharmacists after obtaining informed consent. Study Pharmacists obtain the allocation from the PROSPECT website. Only the Database Manager and Study Pharmacists will have access to the randomization schedule; everyone else remains blinded. Patients receive the intervention until:1) ICU discharge; 2) death; or 3) isolation of Lactobacillus spp. in a sterile site, or if cultured as the sole or predominant organism from a non-sterile site.

RCT Trial Outcomes: The primary outcome is VAP; secondary outcomes include ICU-acquired infections, diarrhea (total, antibiotic-associated and CDAD), antibiotic use, length of stay and mortality in the ICU and hospital, and acquired L. rhamnosus GG infections.

Relevance: Despite clinical uptake of some existing VAP prevention strategies, the morbidity, mortality and cost of VAP underscore the need for further cost-effective interventions to reduce its impact. Whether probiotics impact on VAP, other infections such as CDAD, antibiotic-associated diarrhea or antibiotic use is unclear. When rigorously evaluated, probiotics may have salutary effects decreasing nosocomial infections as prior RCTs suggest; alternatively, probiotics may have no demonstrable effect, or actually cause infections in critically ill patients with impaired immune function.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age
2. Admitted to any ICU and receiving invasive mechanical ventilation
3. Anticipated ventilation of ≥72 hours at the time of screening, as per the ICU physician.

Exclusion Criteria:

1. Invasively mechanically ventilated >72 hours at the time of screening;
2. Patients at potential increased risk of iatrogenic probiotic infection (see Section 2.6 for detailed explanation) including specific immunocompromised populations (HIV <200 CD4 cells/μL, those receiving chronic immunosuppressive medications (e.g., azathioprine, cyclosporine, cyclophosphamide, tacrolimus, methotrexate, mycofenolate, Anti-IL2), previous transplantation (including stem cell) at any time, malignancy requiring chemotherapy in the last 3 months, neutropenia [absolute neutrophil count < 500]). However, patients receiving corticosteroids previously or presently or projected to receive corticosteroids are not excluded;
3. Patients at risk for endovascular infection (previously documented rheumatic heart disease, congenital valve disease, surgically repaired congenital heart disease, unrepaired cyanotic congenital heart disease, any intracardiac repair with prosthetic material [mechanical or bio-prosthetic cardiac valves], previous or current endocarditis, permanent endovascular devices (e.g., endovascular grafts [e.g., aortic aneurysm repair, stents involving large arteries such as aorta, femorals and carotids], inferior vena cava filters, dialysis vascular grafts), tunnelled (not short-term) hemodialysis catheters, pacemakers or defibrillators. Patients with temporary central venous catheters, central venous dialysis catheters or peripherally inserted central catheters (PICCs) are not excluded and patients with coronary artery stents, coronary artery bypass grafts (CABG) or neurovascular coils are not excluded; patients with mitral valve prolapse or bicuspid aortic valve are not excluded providing they have no other exclusion criteria;
4. Patients with a primary diagnosis of severe acute pancreatitis, without reference to a Ranson score [Ranson 1974]). However, patients with mild or moderate pancreatitis are not excluded;
5. Patients with percutaneous gastric or jejunal feeding tubes already in situ as per Health Canada guidance;
6. Strict contraindication or inability to receive enteral medications;
7. Intent to withdraw advanced life support as per the ICU physician;
8. Previous enrolment in this or current enrolment in a potentially confounding tria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2650 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-03-13 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Number of patients with Ventilator Associated Pneumonia (VAP) | 60 Days
  VAP will be diagnosed clinically at each site in patients who are receiving invasive mechanical ventilation for at least 48 hours, when there is a new, progressive or persistent radiographic infiltrate with no other obvious cause and the presence of any 2 of the following symptoms or signs: 1) fever (temperature >38°C) or hypothermia (temperature <36°C as measured by core body temperature); 2) relative neutropenia (<3.0 x 106/L) or leukocytosis (>10 x 106/L) and 3) purulent sputum.

SECONDARY OUTCOMES:
Number of patients with infections acquired during the ICU stay | 60 Days
  Any infection acquired during the ICU stay, defined as respiratory or other infections including bloodstream infections, intravascular catheter-related sepsis, intra-abdominal infections, urosepsis and surgical wound infections.
Number of patients with Clostridium Difficile-associated diarrhea | 60 Days
  3 or more episodes of unformed stools in ≤24 hours and C. difficile toxin positive stool or colonoscopic or histopathologic findings demonstrating pseudomembranous colitis
Number of patients with antibiotic-associated diarrhea | 60 Days
  Antibiotic-associated diarrhea and defined as more than 2 liquid stools a day for 3 or more days in quantities in excess of normal for each patient
Number of patients with diarrhea | 60 Days
  Diarrhea defined as 3 or more loose or watery bowel movements, according to the Bristol Stool Chart (type 6 or 7) and use of a fecal management device
Defined Daily Dose Antibiotic Exposure | 60 Days
  Defined daily dose (DDD), daily doses of therapy (DOT), and antibiotic-free days in ICU
Duration of mechanical ventilation | 60 Days
  Endotracheal tube or tracheostomy, length of ICU stay and length of hospital stay: recorded as number of days
ICU mortality and in-hospital mortality: | 60 Days
  ICU mortality and in-hospital mortality recorded at ICU discharge and hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Cook, MD, Principal Investigator — McMaster University
Locations (44):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
- Canada (41):
  - Peter Louheed Center, Calgary, Alberta
  - Foothills Medical Center, Calgary, Alberta
  - Univeristy of Alberta, Edmonton, Alberta
  - Royal Columbia Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Vancouver, British Columbia
  - Health Science - Winnipeg, Winnipeg, Manatoba
  - St. Boniface, Winnipeg, Manitoba
  - QEII, Halfax, Nova Scotia
  - William Osler Brampton - Brampton Civic Hospital, Brampton, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - Royal Alexandra Hospital, Edmonton, Ontario
  - Hamilton Health Science Centre - Hamilton General Hospital, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Science Centre - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Niagara Health - St. Catharine's Hospital, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - UHN - Toronto Western Hospital, Toronto, Ontario
  - St. Joseph's Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Laval, Quebec
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Center Hospital University Montreal (NCHUM), Montreal, Quebec
  - Center Hospital University Montreal (CHUM) - Notre Dame, Montreal, Quebec
  - Center Hospital University (CHUM) - Saint Luc, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Sacre Coeur Hospital, Montreal, Quebec
  - Hôpital de l'Enfant-Jesus, CHU de Quebec, Québec, Quebec
  - Sherbrooke Hospital, Sherbrooke, Quebec
- King Adulaziz Medical Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Fernando SM, Muscedere J, Rochwerg B, Johnstone J, Daneman N, Marshall JC, Lauzier F, Rudkowski JC, Arabi YM, Heels-Ansdell D, Sligl W, Kristof AS, Duan E, Dionne JC, St-Arnaud C, Reynolds S, Khwaja K, Cook DJ; PROSPECT Investigators and the Canadian Critical Care Trials Group. Frailty and the risk of ICU-acquired infections in a randomised trial: a protocol and statistical analysis plan. BMJ Open. 2025 Nov 13;15(11):e105227. doi: 10.1136/bmjopen-2025-105227. PMID 41248372
- [Derived] Thabane A, Heels-Ansdell D, Zytaruk N, Johnstone J, Lauzier F, Arabi YM, Muscedere J, Clarke F, Hand L, Watpool I, Porteous R, Sandu G, Santos M, Tassy D, Marshall J, McIntyre L, Ball I, Rochwerg B, Karachi T, Zarychanski R, Marquis F, Friedrich JO, Lysecki P, Cook D; PROSPECT Investigators and the Canadian Critical Care Trials Group. Coenrollment of critically ill patients in PROSPECT: characteristics and association with treatment efficacy and safety. Trials. 2025 Sep 26;26(1):370. doi: 10.1186/s13063-025-09028-w. PMID 41013603
- [Derived] Takaoka A, Johnstone J, Lauzier F, Heels-Ansdell D, Davis M, Zytaruk N, Duan E, Dionne J, Saunders L, Arabi YM, Marshall J, Thabane L, Clarke F, Hand L, Masse MH, Rochwerg B, McIntyre L, Girard M, Freitag A, Karachi T, Cook DJ; PROSPECT Investigators; Canadian Critical Care Trials Group. Enrolment patterns in a randomized controlled trial of probiotics in critically ill patients: a retrospective analysis of the PROSPECT trial. Trials. 2024 Dec 27;25(1):851. doi: 10.1186/s13063-024-08701-w. PMID 39731129
- [Derived] Dionne JC, Johnstone J, Heels-Ansdell D, Duan E, Lauzier F, Arabi YM, Adhikari NKJ, Sligl W, Dodek P, Rochwerg B, Marshall JC, Niven DJ, Williamson DR, Reynolds S, Zytaruk N, Cook D. Clostridioides difficile infection in mechanically ventilated critically ill patients: A nested cohort study. J Crit Care. 2023 Jun;75:154254. doi: 10.1016/j.jcrc.2023.154254. Epub 2023 Jan 20. PMID 36682909
- [Derived] Takaoka A, Zytaruk N, Davis M, Matte A, Johnstone J, Lauzier F, Marshall J, Adhikari N, Clarke FJ, Rochwerg B, Lamontagne F, Hand L, Watpool I, Porteous RK, Masse MH, D'Aragon F, Niven D, Heels-Ansdell D, Duan E, Dionne J, English S, St-Arnaud C, Millen T, Cook DJ; PROSPECT Investigators and the Canadian Critical Care Trials Group. Monitoring and auditing protocol adherence, data integrity and ethical conduct of a randomized clinical trial: A case study. J Crit Care. 2022 Oct;71:154094. doi: 10.1016/j.jcrc.2022.154094. Epub 2022 Jun 17. PMID 35724443
- [Derived] Johnstone J, Meade M, Lauzier F, Marshall J, Duan E, Dionne J, Arabi YM, Heels-Ansdell D, Thabane L, Lamarche D, Surette M, Zytaruk N, Mehta S, Dodek P, McIntyre L, English S, Rochwerg B, Karachi T, Henderson W, Wood G, Ovakim D, Herridge M, Granton J, Wilcox ME, Goffi A, Stelfox HT, Niven D, Muscedere J, Lamontagne F, D'Aragon F, St-Arnaud C, Ball I, Nagpal D, Girard M, Aslanian P, Charbonney E, Williamson D, Sligl W, Friedrich J, Adhikari NK, Marquis F, Archambault P, Khwaja K, Kristof A, Kutsogiannis J, Zarychanski R, Paunovic B, Reeve B, Lellouche F, Hosek P, Tsang J, Binnie A, Trop S, Loubani O, Hall R, Cirone R, Reynolds S, Lysecki P, Golan E, Cartin-Ceba R, Taylor R, Cook D; Prevention of Severe Pneumonia and Endotracheal Colonization Trial (PROSPECT) Investigators and the Canadian Critical Care Trials Group. Effect of Probiotics on Incident Ventilator-Associated Pneumonia in Critically Ill Patients: A Randomized Clinical Trial. JAMA. 2021 Sep 21;326(11):1024-1033. doi: 10.1001/jama.2021.13355. PMID 34546300
- [Derived] Johnstone J, Heels-Ansdell D, Thabane L, Meade M, Marshall J, Lauzier F, Duan EH, Zytaruk N, Lamarche D, Surette M, Cook DJ; PROSPECT Investigators and the Canadian Critical Care Trials Group. Evaluating probiotics for the prevention of ventilator-associated pneumonia: a randomised placebo-controlled multicentre trial protocol and statistical analysis plan for PROSPECT. BMJ Open. 2019 Jun 20;9(6):e025228. doi: 10.1136/bmjopen-2018-025228. PMID 31227528